CLINICAL TRIAL: NCT00905307
Title: A Phase 2, 6-Week, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy, Safety, and Tolerability of Oral OPC-34712 Once Daily and Aripiprazole Once Daily for Treatment of Hospitalized Adult Patients With Acute Schizophrenia
Brief Title: Study to Evaluate the Efficacy, Safety, and Tolerability of Oral OPC-34712 and Aripiprazole for Treatment of Acute Schizophrenia
Acronym: STEP 203
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 331-07-203
Record Dates: First submitted 2009-05-19; First posted 2009-05-20 (Estimated); Results first posted 2015-09-03 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-09

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Relapsed
MeSH Terms: conditions — Schizophrenia; Recurrence | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 1 (Experimental): OPC-34712 0.25 mg arm
  Interventions: Drug: OPC-34712
- 2 (Experimental): OPC-34712 low-dose arm
  Interventions: Drug: OPC-34712
- 3 (Experimental): OPC-34712 mid-dose arm
  Interventions: Drug: OPC-34712
- 4 (Experimental): OPC-34712 high-dose arm
  Interventions: Drug: OPC-34712
- 5 (Placebo Comparator)
  Interventions: Drug: Placebo
- 6 (Active Comparator): Aripiprazole arm
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: OPC-34712 — oral, once daily
  Arms: 1; 2; 3; 4
Drug: Placebo — Placebo
  Arms: 5
Drug: Aripiprazole — oral, once daily
  Arms: 6

SUMMARY:
This will be a multicenter, randomized, double-blind, placebo-controlled study designed to assess the tolerability, safety, and efficacy of OPC-34712 (0.25 to 6.0 mg) for the treatment of adult subjects hospitalized with an acute relapse of schizophrenia. Aripiprazole (10 to 20 mg) is included as a positive control to confirm the assay sensitivity of the study. A total of approximately 563 subjects will be screened at an estimated 75 sites worldwide in order to obtain approximately 450 randomized subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between 18 and 65 years of age, with a diagnosis of schizophrenia, as defined by DSM-IV-TR criteria
2. Subjects who have been recently hospitalized or who would benefit from hospitalization for an acute relapse of schizophrenia
3. Subjects experiencing an acute exacerbation of psychotic symptoms

Exclusion Criteria:

1. Females who are breast-feeding and/or who have a positive pregnancy test result prior to receiving study drug
2. Subjects with a current DSM-IV-TR Axis I diagnosis of:

   * Schizoaffective disorder
   * MDD
   * Bipolar disorder
   * Delirium, dementia, amnestic or other cognitive disorder
   * Borderline, paranoid, histrionic, schizotypal, schizoid or antisocial personality disorder
3. Subjects presenting with a first episode of schizophrenia
4. Other protocol specific inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 459 (Actual)
Dates: Start 2009-07; Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (65):
- United States (15):
  - Study Site, Little Rock, Arkansas
  - Study Site, Escondido, California
  - Study Site, Garden Grove, California
  - Study Site, Long Beach, California
  - Study Site, Oceanside, California
  - Study Site, Pasadena, California
  - Study Site, San Diego, California
  - Study Site, Santa Ana, California
  - Study Site, Washington D.C., District of Columbia
  - Study Site, Bradenton, Florida
  - Study Site, Maitland, Florida
  - Study Site, St Louis, Missouri
  - Study Site, Cedarhurst, New York
  - Study Site, Philadelphia, Pennsylvania
  - Study Site, Austin, Texas
- Bulgaria (6):
  - Study Site, Burgas
  - Study Site, Kazanlak
  - Study Site, Pazardzhik
  - Study Site, Plovdiv
  - Study Site, Radnevo
  - Study Site, Rousse
- Croatia (3):
  - Study Site, Rijeka
  - Study Site, Split
  - Study Site, Zagreb
- India (8):
  - Study Site, Vijaywada, Andh Prad
  - Study Site, Visakhapatnam, Andh Prad
  - Study Site, Ahmedabad, Gujarat
  - Study Site, Bangalore, Karna
  - Study Site, Mangalore, Karna
  - Study Site, Pune, Mahara
  - Study Site, Chennai, Tamil Nadu
  - Study Site, Varanasi, Uttar Prad
- Philippines (2):
  - Study Site, Cebu City
  - Study Site, Mandaluyong
- Romania (7):
  - Study Site, Arad
  - Study Site, Bucharest
  - Study Site (1), Bucharest
  - Study Site (2), Bucharest
  - Study Site (3), Bucharest
  - Study Site, Cluj-Napoca
  - Study Site, Oradea
- Russia (3):
  - Study Site, Moscow
  - Study Site, Moscow Region
  - Study Site, Saint Petersburg
- Serbia (4):
  - Study Site (1), Belgrade
  - Study Site (2), Belgrade
  - Study Site, Kragujevac
  - Study Site, Novi Sad
- Slovakia (5):
  - Study Site, Bojnice
  - Study Site, Bratislava
  - Study Site, Liptovský Mikuláš
  - Study Site, Rimavská Sobota
  - Study Site, Žilina
- South Korea (4):
  - Study Site, Busan
  - Study Site, Chuncheon
  - Study Site, Incheon
  - Study Site, Seoul
- Taiwan (2):
  - Study Site, Hualien Town
  - Study Site, Taipei
- Ukraine (6):
  - Study Site, Chernihiv
  - Study Site, Dnipropetrovsk
  - Study Site, Kherson,Vil. Stepanivka
  - Study Site, Kyiv
  - Study Site, Simferopol
  - Study Site, Vinnitsia

REFERENCES:
- [Derived] Kane JM, Skuban A, Hobart M, Ouyang J, Weiller E, Weiss C, Correll CU. Overview of short- and long-term tolerability and safety of brexpiprazole in patients with schizophrenia. Schizophr Res. 2016 Jul;174(1-3):93-98. doi: 10.1016/j.schres.2016.04.013. Epub 2016 May 14. PMID 27188270
- [Derived] Citrome L. Brexpiprazole for schizophrenia and as adjunct for major depressive disorder: a systematic review of the efficacy and safety profile for this newly approved antipsychotic - what is the number needed to treat, number needed to harm and likelihood to be helped or harmed? Int J Clin Pract. 2015 Sep;69(9):978-97. doi: 10.1111/ijcp.12714. Epub 2015 Aug 6. PMID 26250067

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 459 participants recruited at 74 study centres in the United States, Asia and Europe.
  Participants not responding adequately to treatment at Week 4 visit could continue in study and receive open-label OPC-34712 (starting dose 2.5 mg/day with option for decrease to 2 mg/day or increase to 3 mg/day) until Week 6 at study physician's discretion.
Pre-assignment Details: Partipants were randomized in a 1:2:2:2:2:1 ratio to the following groups:
  OPC-34712 0.25 mg arm, OPC-34712 low-dose, OPC-34712 mid-dose, OPC-34712 high-dose, Placebo, Aripiprazole. All other prohibited medications were discontinued at least 24 hours before the first dose of double-blind study medication.
Groups:
- OPC-34712 0.25 mg: 0.25 mg once daily (QD) for 6 weeks
- OPC-34712 Low-dose: 1.0 mg QD starting dose ± 0.5 mg. After a minimum of 2 weeks of treatment, the physician could request a dose increase, if needed for efficacy, based on clinical judgment.
- OPC-34712 Mid-dose: 2.5 mg QD starting dose ± 0.5 mg. After a minimum of 2 weeks of treatment, the physician could request a dose increase, if needed for efficacy, based on clinical judgment.
- OPC-34712 High Dose: 5.0 mg QD starting dose ± 0.5 mg. After a minimum of 2 weeks of treatment, the physician could request a dose increase, if needed for efficacy, based on clinical judgment.
- Aripiprazole: 15 mg QD starting dose ± 5 mg. After a minimum of 2 weeks of treatment, the physician could request a dose increase, if needed for efficacy, based on clinical judgment.
- Placebo: Placebo QD for 6 weeks
Period: Overall Study
Arm/Group | OPC-34712 0.25 mg | OPC-34712 Low-dose | OPC-34712 Mid-dose | OPC-34712 High Dose | Aripiprazole | Placebo
Started | 42 | 89 | 90 | 93 | 50 | 95
Completed | 20 | 52 | 53 | 56 | 34 | 53
Not Completed | 22 | 37 | 37 | 37 | 16 | 42
Not completed — Switched to Open Label Rescue | 7 | 17 | 11 | 11 | 4 | 15
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Adverse Event | 3 | 4 | 5 | 11 | 3 | 5
Not completed — Withdrawal by Subject | 5 | 13 | 15 | 11 | 4 | 13
Not completed — Protocol Violation | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 6 | 3 | 5 | 4 | 4 | 8

BASELINE CHARACTERISTICS:
Groups:
- OPC-34712 0.25 mg: 0.25 mg QD for 6 weeks
- OPC-34712 High-dose: 5.0 mg QD starting dose ± 1.0 mg. After a minimum of 2 weeks of treatment, the physician could request a dose increase, if needed for efficacy, based on clinical judgment.
- Total: Total of all reporting groups
Arm/Group | OPC-34712 0.25 mg | OPC-34712 Low-dose | OPC-34712 Mid-dose | OPC-34712 High-dose | Aripiprazole | Placebo | Total
Number analyzed (Participants) | 42 | 89 | 90 | 93 | 50 | 95 | 459
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.4 (9.1) | 39.2 (10.3) | 37.4 (11.1) | 39.5 (11.1) | 40.8 (11) | 38.8 (11.4) | 39.1 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 36 | 30 | 38 | 16 | 37 | 172
  Male | 27 | 53 | 60 | 55 | 34 | 58 | 287

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 6 in Positive and Negative Syndrome Scale (PANSS) Total Score (Double Blind Phase)
Description: The PANSS consists of three subscales containing a total of 30 symptom constructs. For each symptom construct, severity is rated on a 7-point scale, with a score of 1 indicating absence of symptoms and a score of 7 indicating extremely severe symptoms. PANSS total score is the sum of the rating scores for 7 positive scale items, 7 negative scale items and 16 general psychopathology scale items from the PANSS panel. The PANSS total score ranges from 30-210, with higher scores indicating more severe symptoms.
Time Frame: Baseline to Week 6
Population: Consists of all participants who received at least one dose of study medication and have baseline and at least one post-baseline efficacy evaluation. The last observation carried forward (LOCF) method was used to impute missing data.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- OPC-34712 Mid-dose: 2.5 mg QD starting dose ± 0.5 mg. After a minimum of 2 weeks of treatment , the physician could request a dose increase, if needed for efficacy, based on clinical judgment
Arm/Group | OPC-34712 0.25 mg | OPC-34712 Low-dose | OPC-34712 Mid-dose | OPC-34712 High-dose | Aripiprazole | Placebo
Number analyzed (Participants) | 41 | 88 | 90 | 92 | 50 | 93
Units on a scale | -9.76 (19.29) | -18.73 (20.27) | -16.19 (18.55) | -18.25 (20.49) | -17.98 (21.32) | -14.40 (20.13)
Statistical Analysis 1: Comparison: OPC-34712 Low-dose vs Placebo; Sample size was determined to achieve at least 80% power at alpha level of 0.0167 (two-sided) to detect a difference of -11.5 points in the mean change from baseline in PANSS Total Score at week 6 (LOCF) between an individual OPC-34712 treatment group (except the 0.25 mg QD fixed dose group) and placebo using a two-sided z-test; Test type: Superiority or Other; p = 0.2846, ANCOVA — The Hochberg procedure using two-sided alpha of 0.05 was applied to control the type I error rate at 0.05 level (two-sided) due to multiple comparisons; With treatment and trial center as main effects, and baseline value as covariate; Treatment difference = -4.70, 95% CI 2-sided [-10.2 to 0.82]
Statistical Analysis 2: Comparison: OPC-34712 Mid-dose vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6066, ANCOVA — [p-value comment as in outcome 1, analysis 1]; With treatment and trial center as main effects, and baseline value as covariate; Treatment difference = -1.44, 95% CI 2-sided [-6.96 to 4.07]
Statistical Analysis 3: Comparison: OPC-34712 High-dose vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3293, ANCOVA — [p-value comment as in outcome 1, analysis 1]; With treatment and trial center as main effects, and baseline value as covariate; Treatment difference = -3.86, 95% CI 2-sided [-9.32 to 1.59]
Statistical Analysis 4: Comparison: OPC-34712 0.25 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2263, ANCOVA; With treatment and trial center as main effects, and baseline value as covariate; Treatment difference = 4.62, 95% CI 2-sided [-2.89 to 12.12]
Statistical Analysis 5: Comparison: Aripiprazole vs Placebo; Test type: Superiority or Other; p = 0.3074, ANCOVA; With treatment and trial center as main effects, and baseline value as covariate; Treatment difference = -3.64, 95% CI 2-sided [-10.7 to 3.38]

2. Secondary Outcome: Change From Baseline to Week 6 in PANSS Positive Subscale Score (Double Blind Phase)
Description: The PANSS consists of three subscales containing a total of 30 symptom constructs. For each symptom construct, severity is rated on a 7-point scale, with a score of 1 indicating absence of symptoms and a score of 7 indicating extremely severe symptoms. The positive symptom constructs are delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, and hostility. PANSS positive subscale score is the sum of the rating scores for the 7 positive scale items from the PANSS panel. The PANSS positive subscale score ranges from 7-49, with higher scores indicating more severe symptoms.
Time Frame: Baseline to Week 6
Population: Consists of all participants who received at least one dose of study medication and have baseline and at least one post-baseline efficacy evaluation. The LOCF method was used to impute missing data.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Aripiprazole: 15 mg QD starting dose ± 5 mg.After a minimum of 2 weeks of treatment, the physician could request a dose increase, if needed for efficacy, based on clinical judgment.
Arm/Group | OPC-34712 0.25 mg | OPC-34712 Low-dose | OPC-34712 Mid-dose | OPC-34712 High-dose | Aripiprazole | Placebo
Number analyzed (Participants) | 41 | 88 | 90 | 92 | 50 | 93
Units on a scale | -3.22 (5.26) | -5.97 (7.12) | -4.94 (6.17) | -5.98 (6.72) | -6.60 (7.16) | -4.82 (6.34)
Statistical Analysis 1: Comparison: OPC-34712 0.25 mg vs Placebo; Sample size was determined to achieve at least 80% power at alpha level of 0.0167 (two-sided) to detect a difference of -11.5 points in the mean change from baseline in PANSS positive subscale score at week 6 (LOCF) between an individual OPC-34712 treatment group (except the 0.25 mg QD fixed dose group) and placebo using a two-sided z-test; Test type: Superiority or Other; p = 0.1807, ANCOVA; With treatment and trial center as main effects, and baseline value as covariate; Treatment difference = 1.61, 95% CI 2-sided [-0.75 to 3.97]
Statistical Analysis 2: Comparison: OPC-34712 Low-dose vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1313, ANCOVA; With treatment and trial center as main effects, and baseline value as covariate; Treatment difference = -1.41, 95% CI 2-sided [-3.24 to 0.42]
Statistical Analysis 3: Comparison: OPC-34712 Mid-dose vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.8879, ANCOVA; Treatment difference = -0.13, 95% CI 2-sided [-1.96 to 1.69]
Statistical Analysis 4: Comparison: OPC-34712 High-dose vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1764, ANCOVA; With treatment and trial center as main effects, and baseline value as covariate; Treatment difference = -1.24, 95% CI 2-sided [-3.05 to 0.56]
Statistical Analysis 5: Comparison: Aripiprazole vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1111, ANCOVA; With treatment and trial center as main effects, and baseline value as covariate; Treatment difference = -1.79, 95% CI 2-sided [-4.00 to 0.42]

3. Secondary Outcome: Change From Baseline to Week 6 in PANSS Negative Subscale Score (Double Blind Phase)
Description: The PANSS consists of three subscales containing a total of 30 symptom constructs. For each symptom construct, severity is rated on a 7-point scale, with a score of 1 indicating absence of symptoms and a score of 7 indicating extremely severe symptoms. The 7 negative symptom constructs: blunted affect, emotional withdrawal, poor rapport, passive/apathetic social withdrawal, difficulty in abstract thinking, lack of spontaneity and flow of conversation, stereotyped thinking. PANSS negative subscale score is the sum of the rating scores for the 7 negative scale items from the PANSS panel. The PANSS negative subscale score ranges from 7-49, with higher scores indicating more severe symptoms.
Time Frame: Baseline to Week 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- OPC-34712 0.25 mg: 0.25 mg QD
- OPC-34712 Low-dose: 1.0 mg QD starting dose ± 0.5 mg After a minimum of 2 weeks of treatment (eg, beginning at the Week 2 visit and at any subsequent visit where study medication was dispensed), the investigator could request a dose increase, if needed for efficacy, based on clinical judgment.
- OPC-34712 Mid-dose: 2.5 mg QD starting dose ± 0.5 mg After a minimum of 2 weeks of treatment (eg, beginning at the Week 2 visit and at any subsequent visit where study medication was dispensed), the investigator could request a dose increase, if needed for efficacy, based on clinical judgment.
- OPC-34712 High-dose: 5.0 mg QD starting dose ± 1.0 mg After a minimum of 2 weeks of treatment (eg, beginning at the Week 2 visit and at any subsequent visit where study medication was dispensed), the investigator could request a dose increase, if needed for efficacy, based on clinical judgment.
- Aripiprazole: 15 mg QD starting dose ± 5 mg After a minimum of 2 weeks of treatment (eg, beginning at the Week 2 visit and at any subsequent visit where study medication was dispensed), the investigator could request a dose increase, if needed for efficacy, based on clinical judgment.
- Placebo: Placebo QD
Arm/Group | OPC-34712 0.25 mg | OPC-34712 Low-dose | OPC-34712 Mid-dose | OPC-34712 High-dose | Aripiprazole | Placebo
Number analyzed (Participants) | 42 | 89 | 90 | 93 | 50 | 95
Units on a scale | -1.93 (5.24) | -3.61 (5.15) | -3.84 (5.09) | -3.99 (5.40) | -3.00 (5.74) | -3.17 (4.88)
Statistical Analysis 1: Comparison: OPC-34712 0.25 mg vs Placebo; Sample size was determined to achieve at least 80% power at alpha level of 0.0167 (two-sided) to detect a difference of -11.5 points in the mean change from baseline in PANSS negative subscale score at week 6 (LOCF) between an individual OPC-34712 treatment group (except the 0.25 mg QD fixed dose group) and placebo using a two-sided z-test; Test type: Superiority or Other; p = 0.2896, ANCOVA; With treatment and trial center as main effects, and baseline value as covariate; Treatment difference = 1.00, 95% CI 2-sided [-0.86 to 2.86]
Statistical Analysis 2: Comparison: OPC-34712 Low-dose vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.3701, ANCOVA; With treatment and trial center as main effects, and baseline value as covariate; Treatment difference = -0.61, 95% CI 2-sided [-1.94 to 0.72]
Statistical Analysis 3: Comparison: OPC-34712 Mid-dose vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.6074, ANCOVA; With treatment and trial center as main effects, and baseline value as covariate; Treatment difference = -0.35, 95% CI 2-sided [-1.69 to 0.99]
Statistical Analysis 4: Comparison: OPC-34712 High-dose vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.2777, ANCOVA; With treatment and trial center as main effects, and baseline value as covariate; Treatment difference = -0.73, 95% CI 2-sided [-2.05 to 0.59]
Statistical Analysis 5: Comparison: Aripiprazole vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.8611, ANCOVA; With treatment and trial center as main effects, and baseline value as covariate; Treatment difference = -0.15, 95% CI 2-sided [-1.90 to 1.59]

4. Secondary Outcome: Change From Baseline to Week 6 in Personal and Social Performance Scale (PSP) (Double Blind Phase)
Description: The PSP is a validated clinician-rated scale that measures personal and social functioning in four domains. The rating is based on four main areas: (a) socially useful activities, including work and study; (b) personal and social relationships; (c) self-care; and (d) disturbing and aggressive behaviors. The ratings are converted to a total score based on a 100-point scale using algorithms to identify the appropriate 10-point interval, and the rater's judgment to determine the total score within the 10-point interval. Ratings from 71-100 reflect only mild difficulties. Ratings from 31-70 reflect manifest disabilities of various degrees. Ratings from 1-30 reflect functioning so poor that intensive support or supervision is needed.
Time Frame: Baseline to Week 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OPC-34712 0.25 mg | OPC-34712 Low-dose | OPC-34712 Mid-dose | OPC-34712 High-dose | Aripiprazole | Placebo
Number analyzed (Participants) | 39 | 86 | 84 | 90 | 50 | 90
Units on a scale | 4.54 (13.25) | 11.36 (14.84) | 10.67 (15.21) | 12.17 (14.72) | 10.66 (13.13) | 7.56 (14.90)
Statistical Analysis 1: Comparison: OPC-34712 0.25 mg vs Placebo; Sample size was determined to achieve at least 80% power at alpha level of 0.0167 (two-sided) to detect a difference of -11.5 points in the mean change from baseline in PSP score at week 6 (LOCF) between an individual OPC-34712 treatment group (except the 0.25 mg QD fixed dose group) and placebo using a two-sided z-test; Test type: Superiority or Other; p = 0.3726, ANCOVA; With treatment and trial center as main effects, and baseline value as covariate; Treatment difference = -2.36, 95% CI 2-sided [-7.57 to 2.85]
Statistical Analysis 2: Comparison: OPC-34712 Low-dose vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0664, ANCOVA; With treatment and trial center as main effects, and baseline value as covariate; Treatment difference = 3.80, 95% CI 2-sided [-0.26 to 7.85]
Statistical Analysis 3: Comparison: OPC-34712 Mid-dose vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2944, ANCOVA; With treatment and trial center as main effects, and baseline value as covariate; Treatment difference = 2.20, 95% CI 2-sided [-1.92 to 6.32]
Statistical Analysis 4: Comparison: OPC-34712 High-dose vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0596, ANCOVA; With treatment and trial center as main effects, and baseline value as covariate; Treatment difference = 3.86, 95% CI 2-sided [-0.16 to 7.89]
Statistical Analysis 5: Comparison: Aripiprazole vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1819, ANCOVA; With treatment and trial center as main effects, and baseline value as covariate; Treatment difference = 3.25, 95% CI 2-sided [-1.53 to 8.03]

5. Secondary Outcome: Change From Baseline to Week 6 in Clinical Global Impression-Severity of Illness Scale (CGI-S) Score (Double Blind Phase)
Description: The severity of illness for each participant was rated using the CGI-S. To perform this assessment, the rater or investigator answered the following question: "Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?" Response choices include the following: 0=not assessed; 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients
Time Frame: Baseline to Week 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OPC-34712 0.25 mg | OPC-34712 Low-dose | OPC-34712 Mid-dose | OPC-34712 High-dose | Aripiprazole | Placebo
Number analyzed (Participants) | 41 | 88 | 90 | 92 | 50 | 93
Units on a scale | -0.39 (0.86) | -0.99 (1.29) | -0.87 (1.11) | -1.10 (1.24) | -1.00 (1.21) | -0.82 (1.16)
Statistical Analysis 1: Comparison: OPC-34712 0.25 mg vs Placebo; Sample size was determined to achieve at least 80% power at alpha level of 0.0167 (two-sided) to detect a difference of -11.5 points in the mean change from baseline in CGI-S score at week 6 (LOCF) between an individual OPC-34712 treatment group (except the 0.25 mg QD fixed dose group) and placebo using a two-sided z-test; Test type: Superiority or Other; p = 0.0685, ANCOVA; With treatment and trial center as main effects, and baseline value as covariate; Treatment difference = 0.38, 95% CI 2-sided [-0.03 to 0.79]
Statistical Analysis 2: Comparison: OPC-34712 Low-dose vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0989, ANCOVA; With treatment and trial center as main effects, and baseline value as covariate; Treatment difference = -0.28, 95% CI 2-sided [-0.60 to 0.05]
Statistical Analysis 3: Comparison: OPC-34712 Mid-dose vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8006, ANCOVA; With treatment and trial center as main effects, and baseline value as covariate; Treatment difference = -0.04, 95% CI 2-sided [-0.37 to 0.28]
Statistical Analysis 4: Comparison: OPC-34712 High-dose vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0898, ANCOVA; With treatment and trial center as main effects, and baseline value as covariate; Treatment difference = -0.28, 95% CI 2-sided [-0.60 to 0.04]
Statistical Analysis 5: Comparison: Aripiprazole vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2851, ANCOVA; With treatment and trial center as main effects, and baseline value as covariate; Treatment difference = -0.21, 95% CI 2-sided [-0.59 to 0.18]

6. Secondary Outcome: Mean Clinical Global Impression - Improvement (CGI-I) at Week 6
Description: The rater or investigator rated the particpant's total improvement whether or not it was due entirely to drug treatment. All responses were compared to the participant's condition at baseline prior to the first dose of double-blind study medication. Response choices included the following: 0=not assessed; 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; 7=very much worse.
Time Frame: Week 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | OPC-34712 0.25 mg | OPC-34712 Low-dose | OPC-34712 Mid-dose | OPC-34712 High-dose | Aripiprazole | Placebo
Number analyzed (Participants) | 41 | 88 | 90 | 92 | 50 | 93
Units on a scale | 3.66 (1.48) | 3.08 (1.58) | 3.17 (1.45) | 3.04 (1.50) | 3.04 (1.52) | 3.34 (1.54)
Statistical Analysis 1: Comparison: OPC-34712 0.25 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4008, Cochran-Mantel-Haenszel; The Cochran-Mantel-Haenszel (CMH) row mean scores differ test controlling for study center was applied to mean CGI-I score
Statistical Analysis 2: Comparison: OPC-34712 Low-dose vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1117, Cochran-Mantel-Haenszel; The CMH row mean scores differ test controlling for study center was applied to mean CGI-I score
Statistical Analysis 3: Comparison: OPC-34712 Mid-dose vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2739, Cochran-Mantel-Haenszel; The CMH row mean scores differ test controlling for study center was applied to mean CGI-I score
Statistical Analysis 4: Comparison: OPC-34712 High-dose vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1045, Cochran-Mantel-Haenszel; The CMH row mean scores differ test controlling for study center was applied to mean CGI-I score
Statistical Analysis 5: Comparison: Aripiprazole vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1149, Cochran-Mantel-Haenszel; The CMH row mean scores differ test controlling for study center was applied to mean CGI-I score

7. Secondary Outcome: Response Rate at Week 6
Description: Response rate was defined as a reduction of ≥ 30% from baseline in PANSS Total Score; or a CGI-I score of 1 (very much improved) or 2 (much improved) at Week 6
Time Frame: Week 6
Population: Consists of all participants who received at least one dose of study medication and have baseline and at least one post-baseline efficacy evaluation. The LOCF method was used to impuite missing data.
Measure: Number; unit: Percentage of participants
Groups:
- OPC-34712 High-dose: 5.0 mg QD starting dose ± 1.0 mg. After a minimum of 2 weeks of treatment, the investigator could request a dose increase, if needed for efficacy, based on clinical judgment.
Arm/Group | OPC-34712 0.25 mg | OPC-34712 Low-dose | OPC-34712 Mid-dose | OPC-34712 High-dose | Aripiprazole | Placebo
Number analyzed (Participants) | 42 | 89 | 90 | 93 | 50 | 95
Percentage of participants | 40.5 | 57.3 | 46.7 | 51.6 | 60.0 | 49.5
Statistical Analysis 1: Comparison: OPC-34712 0.25 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6200, Cochran-Mantel-Haenszel; CMH general association test controlling for study center will be applied to the analysis of response rate; Relative Risk = 0.89, 95% CI 2-sided [0.57 to 1.40]
Statistical Analysis 2: Comparison: OPC-34712 Low-dose vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1501, Cochran-Mantel-Haenszel; CMH general association test controlling for study center will be applied to the analysis of response rate; Relative Risk = 1.19, 95% CI 2-sided [0.95 to 1.48]
Statistical Analysis 3: Comparison: OPC-34712 Mid-dose vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5271, Cochran-Mantel-Haenszel; CMH general association test controlling for study center will be applied to the analysis of response rate; Relative Risk = 0.91, 95% CI 2-sided [0.66 to 1.25]
Statistical Analysis 4: Comparison: OPC-34712 High-dose vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8670, Cochran-Mantel-Haenszel; CMH general association test controlling for study center will be applied to the analysis of response rate; Relative Risk = 1.02, 95% CI 2-sided [0.78 to 1.34]
Statistical Analysis 5: Comparison: Aripiprazole vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3892, Cochran-Mantel-Haenszel; CMH general association test controlling for study center will be applied to the analysis of response rate; Relative Risk = 1.15, 95% CI 2-sided [0.85 to 1.56]

8. Secondary Outcome: Discontinuation Rate for Lack of Efficacy or Receipt of Open Label OPC-34712
Description: Efficacy-related discontinuation rate was assessed
Time Frame: Baseline to Week 6
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Groups:
- OPC-34712 Low-dose: 1.0 mg QD starting dose ± 0.5 mg. After a minimum of 2 weeks of treatment, the physicna could request a dose increase, if needed for efficacy, based on clinical judgment.
Arm/Group | OPC-34712 0.25 mg | OPC-34712 Low-dose | OPC-34712 Mid-dose | OPC-34712 High-dose | Aripiprazole | Placebo
Number analyzed (Participants) | 42 | 89 | 90 | 93 | 50 | 95
Percentage of participants | 31 | 22.5 | 17.8 | 16.1 | 16.0 | 24.2
Statistical Analysis 1: Comparison: OPC-34712 0.25 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8540, Cochran-Mantel-Haenszel — Derived using CMH test stratified by trial center; Relative risk = 1.06, 95% CI 2-sided [0.59 to 1.88]
Statistical Analysis 2: Comparison: OPC-34712 Low-dose vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4492, Cochran-Mantel-Haenszel — Derived using CMH test stratified by trial center; Relative Risk = 0.82, 95% CI 2-sided [0.49 to 1.38]
Statistical Analysis 3: Comparison: OPC-34712 Mid-dose vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1854, Cochran-Mantel-Haenszel — Derived using CMH test stratified by trial center; Relative Risk = 0.67, 95% CI 2-sided [0.36 to 1.23]
Statistical Analysis 4: Comparison: OPC-34712 High-dose vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0946, Cochran-Mantel-Haenszel — Derived using CMH test stratified by trial center; Relative Risk = 0.61, 95% CI 2-sided [0.33 to 1.10]
Statistical Analysis 5: Comparison: Aripiprazole vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2133, Cochran-Mantel-Haenszel — Derived using CMH test stratified by trial center; Relative Risk = 0.63, 95% CI [0.30 to 1.34]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were recorded from the time of signing the informed consent, during the 6-week treatment period and up to 30 days after the last dose of study medication. The AEs presented are for the double blind phase.
Arm/Group | OPC-34712 0.25 mg | OPC-34712 Low-dose | OPC-34712 Mid-dose | OPC-34712 High-dose | Aripiprazole | Placebo
Serious Adverse Events (participants affected / at risk) | 0/42 | 3/89 | 5/90 | 4/93 | 2/50 | 3/95
Other Adverse Events (participants affected / at risk) | 20/42 | 41/89 | 36/90 | 52/93 | 22/50 | 39/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OPC-34712 0.25 mg (N=42) | OPC-34712 Low-dose (N=89) | OPC-34712 Mid-dose (N=90) | OPC-34712 High-dose (N=93) | Aripiprazole (N=50) | Placebo (N=95)
Death (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1 | 0
Complex partial seizures (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1
Schizophrenia (Psychiatric disorders) | 0 | 1 | 1 | 1 | 0 | 1
Schizophrenia, paranoid type (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OPC-34712 0.25 mg (N=42) | OPC-34712 Low-dose (N=89) | OPC-34712 Mid-dose (N=90) | OPC-34712 High-dose (N=93) | Aripiprazole (N=50) | Placebo (N=95)
Diarrhoea (Gastrointestinal disorders) | 3 | 5 | 1 | 4 | 4 | 3
Dyspepsia (Gastrointestinal disorders) | 4 | 4 | 3 | 4 | 1 | 7
Nausea (Gastrointestinal disorders) | 1 | 4 | 7 | 6 | 1 | 2
Vomiting (Gastrointestinal disorders) | 2 | 2 | 6 | 2 | 3 | 6
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 2 | 5 | 0 | 1
Weight increased (Investigations) | 1 | 6 | 9 | 6 | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 3 | 3 | 0 | 1
Akathisia (Nervous system disorders) | 1 | 6 | 5 | 14 | 2 | 4
Dizziness (Nervous system disorders) | 0 | 4 | 2 | 5 | 1 | 3
Extrapyramidal disorder (Nervous system disorders) | 0 | 3 | 3 | 6 | 2 | 4
Headache (Nervous system disorders) | 6 | 8 | 13 | 7 | 3 | 10
Somnolence (Nervous system disorders) | 0 | 3 | 3 | 5 | 0 | 2
Agitation (Psychiatric disorders) | 4 | 4 | 4 | 7 | 5 | 4
Anxiety (Psychiatric disorders) | 5 | 7 | 6 | 10 | 5 | 10
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 2 | 3 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 4 | 2 | 6 | 1 | 8
Insomnia (Psychiatric disorders) | 4 | 12 | 9 | 9 | 4 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No